CLINICAL TRIAL: NCT00568724
Title: Urinary Biomarkers as Predictors on Renal Function in Congenital Hydronephrosis
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MGM-01
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Ureteral Obstruction
Keywords: Hydronephrosis; Ureteral obstruction
MeSH Terms: conditions — Ureteral Obstruction; Hydronephrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine and frozen pelvic tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Children referred to surgical treatment of congenital hydronephrosis
- 2: 15 age- and sex-matched controls
- Children with healthy pelvic tissue: Children referred to nephrectomy due to nephrotic syndrome
- Adults with healthy pelvic tissue: Adults referred to nephrectomy due to another cause than hydronephrosis

SUMMARY:
The purpose of this study is to detect new urinary biomarkers that can be used as predictors on renal function in congenital hydronephrosis caused by unilateral ureteral obstruction (UUO) and to elucidate the pathophysiology of UUO.

ELIGIBILITY:
Inclusion Criteria:

* Children referred to surgical treatment of congenital hydronephrosis caused by ureteral obstruction.
* Declining function of the hydronephrotic kidney more than 5 %, and to less than 40 % of the total renal function OR ipsilateral flank pain.

Exclusion Criteria:

* Bilateral hydronephrosis
* Previous operation in the urinary system except operation for phimosis and other deformations of the external genital organs.
* Deformations in the lower part of the ureter, bladder and urethra. Urinary stones. Reflux. Urinary tract infections < 6 months.
* Neurogenic bladder dysfunction.
* GFR < 40 % standardized to age.
* Non-compliance. Linguistic difficulties.

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children referred to surgical treatment of congenital hydronephrosis caused by ureteral obstruction.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2007-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Urinary cytokines | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Troels M Jørgensen, Professor, MD, Principal Investigator — Department of Urology, Aarhus University Hospital Skejby
Locations (1):
- Institute of Clinical Medicine, University of Aarhus, Aarhus, Denmark

REFERENCES:
- [Background] Madsen MG, Norregaard R, Palmfeldt J, Olsen LH, Frokiaer J, Jorgensen TM. Urinary NGAL, cystatin C, beta2-microglobulin, and osteopontin significance in hydronephrotic children. Pediatr Nephrol. 2012 Nov;27(11):2099-2106. doi: 10.1007/s00467-012-2217-6. Epub 2012 Jun 19. PMID 22710694